CLINICAL TRIAL: NCT01714986
Title: Psychological Impact, Metabolic Control, Biological Stress Markers in Diabetes: Intervention With Affect School and Basal Body Awareness
Brief Title: Psychological Variables and Hyperglycemia in Diabetes Mellitus
Acronym: ALEXIDIAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not active
Sponsor: Lund University (Other)
Collaborators: FoU Kronoberg, Landstinget Kronoberg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FoU-Kronoberg 4522
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus; Depression; Alexithymia; Anxiety
Keywords: Diabetes mellitus; Depression; Anxiety; Alexithymia; Self Image; HbA1c; Psychoeducation
MeSH Terms: conditions — Diabetes Mellitus; Depression; Affective Symptoms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Affect School (Active Comparator): Psychological group education intervention
  Interventions: Behavioral: Affect School
- Body Awareness Therapy (Active Comparator): Physiotherapeutic psychosomatic intervention
  Interventions: Behavioral: Body Awareness Therapy

INTERVENTIONS:
Behavioral: Affect School
  Arms: Affect School
Behavioral: Body Awareness Therapy
  Arms: Body Awareness Therapy

SUMMARY:
The investigators want to try the psycho educational method "The Affect School with Script Analysis and the physiotherapeutic mind-body therapy "Basal Body Awareness Therapy in patients with diabetes, high HbA1c and psychological symptoms, in order to improve psychological health- with the primary outcome reduced depression. Secondary outcomes are improved improved glycemic control and self-image, and reduced alexithymia and anxiety.

DETAILED DESCRIPTION:
Background:

Depression is common in patients with diabetes and is associated with impaired glycemic control and elevated cortisol levels. Alexithymia has been associated with depression, anxiety, stress related disorders and diabetes mellitus. Affect School (AS) is an intervention that may reduce depression and alexithymia according to previous research. Basic Body Awareness Therapy (BBAT) is a stress-reducing technique and is used in psychiatric care in Scandinavia in order to improve psychiatric health.

Purpose:

The aims are to: 1. Analyze the prevalence of depression and anxiety and the personality variables alexithymia and self image in diabetes patients at baseline. 2. Explore correlations between these variables and risk factors, including biochemical markers for diabetic complications. 3. To evaluate an intervention with Affect School with Script Analysis and Basal Body Awareness Therapy in patients with diabetes that scored high in psychometric self-report tests and at the same time showed impaired metabolic control.

Method:

A randomized controlled trial in two steps. First step started in 2009 and consists of 350 people with diabetes, 90% with type 1 diabetes, 18-59 years, 56% men, 44% women. Base-line study: from medical records and the National Diabetes Registry - waist circumference, BMI, blood pressure, type and duration of diabetes, diabetes complications, other diseases, medications, exercise habits and smoking. Tests - A1c, blood lipids, cytokines, hormones, beta-cell antibodies, c-peptide, midnight cortisol (salivary). Self-report tests of psychological and personality variables: HAD, TAS-20, SASB. Intervention: patients with HbA1c >70 mmol/mol (A1c ≥ 8 %) and anxiety (HAD ≥ 8), depression (HAD ≥ 8), negative self-image (SASB: Affinity dimension <284) or alexithymia (TAS-20 ≥ 61) were randomized to AS or BBA. AS: 8 group sessions followed by 10 individual sessions. Instructors were a primary care physician and a psychotherapist. BBA: 10 group meetings and 5individual sessions with a physiotherapist as instructor. Post intervention: Self report tests, A1c, cortisol.

Second step will start in 2015: Recruitment of 350 people from primary care with type 2 diabetes with high A1c and either depression, alexithymia, negative self image or anxiety. Randomization procedures and patient characteristics will be assessed in the same way as above.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes and diabetes duration ≥1 year and HbA1c >70 mmol/mol, and one of the following: depression, alexithymia, anxiety or a negative self image.

Exclusion Criteria:

•1) pregnancy; 2) severe comorbidities if it is anticipated that participation will be difficult or unsafe for the patient (end-stage renal disease, cancer, hepatic failure, deafness, social blindness, psychotic disorder, bipolar disorder, suicide ideation, severe personality disorder or severe substance abuse), 3) cognitive deficiencies (mental retardation, stroke or dementia); or 5) inadequate Swedish

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intervention with Affect School with Script Analysis and Basic Basal Awareness Therapy in patients with diabetes, psychological symptoms and high HbA1c | First follow up after intervention about 2 years after baseline and terminal follow up 6 years from baseline
  a two-arm randomized controlled trial comparing Affect School and Basal Body Awareness Therapy

SECONDARY OUTCOMES:
Level of HbA1c | First follow up after intervention about 2 years after baseline and terminal follow up 6 years from baseline
  Compare the HbA1c level before and after intervention
Alexithymia | First follow up after intervention about 2 years after baseline and terminal follow up 6 years from baseline
  Includes difficulty identifying and describing feelings and low capacity of introspection and reflection - assessed by Toronto Alexithymia Scale 20-items
Anxiety | First follow up after intervention about 2 years after baseline and terminal follow up 6 years from baseline
  Assessed by Hospital Anxiety and Depression scale -Anxiety subscale (HADS-a)
Self-image | First follow up after intervention about 2 years after baseline and terminal follow up 6 years from baseline
  Assessed by Structural Analysis of Social Behaviour -Affinity dimension (SASB - Aff)

CONTACTS AND LOCATIONS:
Overall Officials: Eva O Melin, MD, Principal Investigator — Fou Kronoberg, Kronoberg County Council, Växjö, Sweden

REFERENCES:
- [Derived] Melin EO, Svensson R, Gustavsson SA, Winberg A, Denward-Olah E, Landin-Olsson M, Thulesius HO. Affect school and script analysis versus basic body awareness therapy in the treatment of psychological symptoms in patients with diabetes and high HbA1c concentrations: two study protocols for two randomized controlled trials. Trials. 2016 Apr 27;17(1):221. doi: 10.1186/s13063-016-1347-8. PMID 27121185